CLINICAL TRIAL: NCT06643715
Title: Research of the Application of Pancreatic Cancer Screening Artificial Intelligence Model 'PANDAPro': A Single-Center,Realworld Clinical Trial
Brief Title: Research of the Application of Pancreatic Cancer Screening Artificial Intelligence Model "PANDAPro"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Lishui Municipal Central Hospital (Other Government); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZY-PANDAPro
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: Artificial Intelligence; Pancreatic Cancer; PANDA PLUS; PANDA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The PANDA (Pancreatic Cancer Detection with Artificial Intelligence) early screening model was developed by Alibaba DAMO Academy.It employs a fully automated pancreatic segmentation model using the VoxelMorph algorithm, which enhances registration speed and accuracy. By building a self-learning framework, the model efficiently obtains precise annotations of non-contrast CT images. The core network is based on Transformer technology, combined with the MaskFormer model to improve diagnostic accuracy.
  The upgraded PANDA Pro model has improved upon the original PANDA model by enhancing its ability to differentiate between pancreatitis, pancreatic cystic lesions, and eliminating interference from adjacent organs such as the common bile duct and duodenum. These advancements have effectively increased the model's clinical utility, making it more reliable for real-world applications in diagnosing pancreatic conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PANDA Pro (Experimental): recall of clinically missed but PANDA Pro detected pancreatic lesions
  Interventions: Device: PANDA Pro

INTERVENTIONS:
Device: PANDA Pro — Patients with PANDA Pro-reported PDAC positivity but no pancreatic lesions indicated in the imaging report, or those with positive pancreatic findings in the imaging report but no subsequent clinical intervention, will be identified as requiring follow-up. These patients will be recalled to the First Affiliated Hospital of Zhejiang University for further examination and diagnosis.

SUMMARY:
The purpose of this study is to build upon the previously developed deep learning-based non-contrast CT pancreatic cancer screening model, PANDA. The model will first undergo training and enhancement, followed by external validation across multiple centers. Subsequently, a large-scale real-world validation will be conducted at Zhejiang University's First Affiliated Hospital , the study will be divided into two rounds. In the first round, the performance of the PANDA model and the upgraded PANDA Pro model will be compared on consecutive retrospective real-world CT scans. In the second round, physicians will record the PANDA Pro results in real time to identify potential pancreatic lesions that may have been clinically missed. By leveraging clinical big data across different scenarios at Zhejiang University's First Affiliated Hospital, the study aims to validate the model's role in prompting and supplementing the diagnosis of PDAC in clinical practice, thereby laying the foundation for large-scale opportunistic screening of PDAC.

DETAILED DESCRIPTION:
In the first round of real-world validation, abdominal enhanced CT imaging data from patients treated at the First Affiliated Hospital of Zhejiang University between January 2018 and July 2022 were consecutively included. The results of both PANDA and PANDA Pro were recorded and compared with the pathological gold standard of the patients to evaluate model performance.

In the second round of real-world validation, patients with non-contrast CT scans from November 1st, 2025, to August 1, 2027, are expected to be enrolled. The enrolled patients will be categorized into three groups: nonPDAC, PDAC, and normal. The results will be compared with imaging report findings. Patients with PANDA Pro-reported PDAC positivity but no pancreatic lesions indicated in the imaging report, or those with positive pancreatic findings in the imaging report but no subsequent clinical intervention, will be identified as requiring follow-up. These patients will be recalled to the First Affiliated Hospital of Zhejiang University for further examination and diagnosis. Among them, patients with secondary examination confirming PDAC positivity will undergo standard clinical procedures such as MDT at the hospital, ultimately tracking their treatment to confirm ground truth. For patients with secondary examination indicating PDAC negativity, a preliminary determination of their true status will be made after a small-scale discussion between hepatobiliary surgeons and radiologists. Those judged as false positives will undergo follow-up for up to two years to determine their outcomes, thereby validating the sensitivity and specificity of the PANDA Pro model. For patients with PANDA Pro-reported nonPDAC positivity but no positive pancreatic findings in the imaging report, hepatobiliary-pancreatic surgeons and radiologists will retrospectively review the images to confirm their true status. For patients with PANDA Pro-reported normal results but imaging reports indicating pancreatic lesions, a secondary review by surgeons will be conducted to determine whether it is a false negative by PANDA Pro.

For patients reported as true positives for PDAC by the PANDA Pro model, medical records (including tumor marker levels, patient symptoms, resectability classification, TNM staging, etc.) will be collected. These will be compared with corresponding indicators from PDAC patients identified through the SOC(Standard Order of Clinic) during the same period, to validate PANDA Pro's ability to detect and identify lesions in the early stages of pancreatic cancer development.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone chest and/or abdominal CT scans at outpatient clinics, inpatient departments, or physical examination centers;
* Age at the time of the scan between 18-90 years old, with no restriction on gender;

Exclusion Criteria:

* Chest CT scans that do not cover the pancreas;
* Non-contrast CT scans performed in emergency settings;
* Patients who have undergone thoracic/abdominal surgeries affecting or altering the anatomical display of the pancreas (e.g., post-esophageal, gastric, pancreatic, vascular surgeries, or post-ERCP);
* Non-standard scans (e.g., hands placed on either side of the body or abdomen, severe respiratory motion artifacts, perfusion contamination, etc.);
* CT scans ordered by hepatobiliary and pancreatic surgeons or oncologists;
* Patients referred to a higher-level hospital due to a pancreatic mass found during local hospital examination;
* Patients who, for personal reasons, did not follow up with pancreatic cancer diagnosis or treatment at the hospital, or were lost to follow-up midway;
* Patients with concurrent malignancies in other locations or those undergoing comprehensive cancer treatment for malignant tumors;
* Imaging reports made by radiologists without referring to AI during the image interpretation;
* Patients who underwent enhanced CT, MRI, or PET-CT examinations concurrently.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection efficiency of doctors in pancreatic cancer assisted by PANDA Pro | Complete the statistics within six months after the patient is fully enrolled, and it is expected to take 2 years from the start of the study
  Sensitivity、Specificity、PPV、NPV

SECONDARY OUTCOMES:
TNM stage | 1 day (evaluate through CT imaging before surgery)
  Staging of pancreatic cancer
Resectability grading | 1 day (evaluate through CT imaging before surgery)
  Resectability grading of pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No